CLINICAL TRIAL: NCT00695968
Title: A Prospective Study Evaluating Breast Density and the Role of Preoperative Mammography, Ultrasound, Elastography, and Magnetic Resonance Imaging in the Detection of Breast Cancer
Brief Title: Breast Density and the Role of Preoperative Mammography, Ultrasound, Elastography and MRI
Status: Terminated | Type: Observational
Why Stopped: low accrual
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: BRSNSTU0024; 98159 (Other: SU); BRSNSTU0024
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2012-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To determine the sensitivity, specificity, and accuracy of preoperative ultrasound, elastography, mammography and breast MRI in women with dense breast tissue diagnosed with breast cancer; to test whether elastography or MRI can improve upon routine mammogram and conventional ultrasound in women with dense breast tissue.

ELIGIBILITY:
Inclusion Criteria:- Patients must have a suspicious breast lesion detected by a physical exam, mammography or U/S . that has not been surgically resected and is being considered to undergo biopsy if clinically indicated.

* Patients must be >= 18 and < 80 years of age, and female.
* Patients must have the ability to understand and the willingness to sign a written informed consent document. Exclusion Criteria:- Patients who have already had primary surgical excision of the suspicious finding
* <18 or >80 years of age
* Pregnant or Lactating Women

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must have a suspicious breast lesion
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2008-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra M Ikeda, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States